CLINICAL TRIAL: NCT05639647
Title: A PHASE 2A MULTICENTER, OBSERVER-BLINDED, RANDOMIZED 2 ARM STUDY TO INVESTIGATE PHARMACOKINETICS, SAFETY, TOLERABILITY AND EFFICACY OF INTRAVENOUS AZTREONAM-AVIBACTAM ± METRONIDAZOLE COMPARED TO BEST AVAILABLE THERAPY (BAT) IN PEDIATRIC PARTICIPANTS 9 MONTHS TO LESS THAN 18 YEARS OF AGE WITH SERIOUS GRAM-NEGATIVE BACTERIAL INFECTIONS INCLUDING COMPLICATED INTRA-ABDOMINAL INFECTION
Brief Title: Study of 2 Medicines (Aztreonam and Avibactam) Compared to Best Available Therapy for Serious Gram-negative Infections
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C3601008; 2022-501575-12-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-10-24; First posted 2022-12-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Gram-negative Bacterial Infections
Keywords: Gram-negative bacterial infections
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — Aztreonam; avibactam

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, parallel study comparing ATM-AVI with or without metronidazole (MTZ) compared to BAT for the treatment of serious gram-negative bacterial infections. For every 3 participants assigned to ATM-AVI therapy one will be assigned to BAT.
Who Masked: Investigator
Masking Description: Blinded observer assigned by each site
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATM-AVI (Experimental): ATM-AVI administered iv every 6 or 8 hours and dosed according to participant's weight and kidney function for up to 14 days depending on response. At the investigator's discretion, the participant may be switched to oral therapy after 3 days of iv ATM-AVI therapy
  Interventions: Drug: ATM-AVI
- Best available therapy (BAT) (Active Comparator): BAT will be selected by the investigator and administered iv. At the investigator's discretion, the participant may be switched to oral therapy after 3 days of iv BAT
  Interventions: Drug: BAT

INTERVENTIONS:
Drug: ATM-AVI — A drug specifically designed to treat resistant gam-negative bacterial infections
  Other Names: aztreonam plus avibactam
  Arms: ATM-AVI
Drug: BAT — BAT will be selected by the investigator and administered iv as appropriate for the selected drug(s)
  Other Names: Best available therapy
  Arms: Best available therapy (BAT)

SUMMARY:
The purpose of this study is to evaluate how Aztreonam (ATM) and Avibactam (AVI) are processed in pediatric participants. This study also aims to understand participant safety and effects in pediatric participants.

The study is seeking participants who are:

* 9 months to less than 18 years of age
* Hospitalized
* Suspected/known to have a gram-negative infection
* Receiving intravenous (iv, given directly into a vein) antibiotics
* Being treated for complicated infections of various body parts that includes the abdomen, urinary tract, blood stream, and lungs.
* Participants will receive either ATM-AVI or best available therapy (BAT).
* Both therapies will be given through a vein.
* Participants with complicated abdominal infections will also receive iv Metronidazole (MTZ). Patients with cIAI and Cockayne Syndrome are excluded due to a risk of severe hepatotoxicity with the use of MTZ. - Participants on ATM-AVI treatment who have anaerobic infections will also receive iv MTZ at the study doctor's discretion.
* The iv dose of ATM-AVI will be based on the participant's weight and kidney function.
* The study doctor will determine the iv dose of BAT.
* During the first 2 study days, participants on ATM-AVI therapy will have 5 blood draws in small quantities.
* Starting on day 4, the study doctor will decide if participants may be switched to oral therapy.
* Participants will receive a maximum of 14 days of ATM-AVI treatment.
* After discharge from the hospital, 1 study visit may be required.
* Depending on the participant's response, the study duration will be from 33 to 50 days.
* The investigator will contact participants by phone 28 to 35 days after the last study treatment to check participants health status.

DETAILED DESCRIPTION:
* Following informed consent, potential participants who are hospitalized, receiving IV antibiotics for less than 24 hours within 48 hours of randomization or failed antibiotic therapy for greater than 48 hours and have suspected/known gram-negative bacterial infections with a complex intra-abdominal infection (cIAI), complex urinary tract (cUTI), blood stream infection (BSI), hospital acquired pneumonia or ventilator associated pneumonia (HAP/VAP) will be screened.
* Although cultures are required, isolation of the causative pathogen is not a criteria for enrollment. - cUTI participants requiring systemic prophylactic antibiotics for any reason at screening are allowed to enter the study provided they discontinue this medication prior to first study drug dose.
* If the participant satisfies the inclusion and exclusion requirements, the participant will be randomly enrolled in a ratio of 3 iv ATM-AVI for each iv BAT.
* A total of 48 participants at approximately 33 sites will be randomized using interactive response technology (IRT).
* The study will be multicenter, international and open label with a single blinded observer assigned by each investigational site.
* There will be 4 cohorts with ages 12 to less than 18 years (Cohort 1), 6 to less than 12 years (Cohort 2), 2 to less than 6 years (Cohort 3) and 9 months to less than 2 years (Cohort 4).
* Each cohort will have 12 participants for a total of 48 participants.
* Cohorts 1 and 2 will be enrolled simultaneously. - - Cohort 3 will begin enrollment after the first 4 participants complete Cohort 2 and PK data and safety have been reviewed by the sponsor and an external data monitoring committee (DMC). Then ATM-AVI dose may be adjusted as needed.
* Cohort 4 will begin enrollment after the first 4 participants completed Cohort 3 and the PK data have been reviewed by the sponsor and the DMC. Then the ATM-AVI dose may be adjusted as needed.
* After 4 participants complete Cohort 4 the PK data will be review by the sponsor and DMC and then the ATM-AVI dose may be adjusted as needed.
* Enrollment will not be paused during the PK data reviews of the first 4 ATM-AVI participants in a cohort. If the ATM-AVI dose requires adjustment, the cohort 4 number will be increased to 20 with 15 receiving ATM-AVI and 5 BAT.
* All participants in the ATM-AVI group will receive an initial ATM-AVI loading dose and then maintenance doses every 6 or 8 hours depending on the participant's weight and kidney function.
* ATM-AVI will be infused over 3 hours.
* Those with cIAI will receive metronidazole (MTZ). Patients with cIAI and Cockayne Syndrome are excluded due to a risk of severe hepatotoxicity with the use of MTZ. - At the investigator's discretion MTZ will be administered to those with BSI, cUTI or HAP/VAP and an associated anaerobic infection.
* MTZ will be administered iv over 20 to 30 minutes starting.
* Optional gram-positive coverage with vancomycin, teicoplanin and linezolid is permitted. Daptomycin is only permitted for cIAI and BSI participants.
* Coverage with iv aminoglycoside is permitted for Pseudomonas aeruginosa.
* Concerning concomitant medications, participants with cUTI may not take prophylactic therapy during study drug treatment.
* Systemic antibiotics are not permitted unless the study drug failed, or it is for a remote site infection essential for participant's safety.
* Systemic iv antivirals are permitted.
* Systemic antifungals should be avoided unless indicated.
* Meropenem/carbapenem-type antibiotics cannot be given concomitantly with ATM-AVI.
* Probenecid and inhaled antibiotics are to be avoided from informed consent until the end of iv treatment (EOIV).
* Antibiotic peritoneal lavage is not permitted. Non-antibiotic lavage is permitted.
* The primary endpoints are pharmacokinetics (PK) and safety.
* Five PK micro-blood samples of at least 0.1 mL will be drawn. The initial 2 PK micro blood samples will be drawn at 2 hours and 5 hours after the first infusion. The next 3 PK micro-blood samples will be drawn at 15 minutes before, 5 hours and 5 3/4 hours after the 5th infusion or a later infusion.
* ATM and AVI clearance (CL), maximum (Cmax) and minimum (Cmin) venous blood concentration, area under the curve (AUC) and half-life (t1/2) will be analyzed.
* A blinded observer (BO), assigned by each investigational site, will clinically assess the participants every day.
* The BO will evaluate causality of all adverse events (AEs) and serious adverse events (SAEs) while the participant is in the hospital, within 24 hours of the end of iv study drug (EOIV), and within 48 hours of end of treatment for those switched to oral therapy.
* For the secondary endpoint of efficacy, the BO will clinically assess the test of cure (TOC) within 7 to 14 days of the last antibiotic treatment. Potential for liver function abnormalities and acute kidney injury will be specifically monitored in addition to standard of care assessments.
* Cure is defined as signs and symptoms improved with no further antimicrobial treatment required except for adjunctive gram-positive therapy or for Pseudomonas aeruginosa.
* In addition, for cIAI participants, no unplanned drainage or surgical intervention is necessary since the initial surgical procedure. Only for those switched to oral therapy before 14 days, improvement is afebrile with absence of new signs or symptoms and improvement of 1 or more symptoms or signs with no worsening of signs or symptoms.
* Failure is defined as death, requirement of antibiotics for the index infection, or discontinuation due to an AE(s). cIAI participants have additional failure criteria of requiring surgical intervention and/or have an infected post-surgical wound(s).
* Participant may choose to permanently discontinue and are free to discontinue treatment without further treatment prejudice. Possible reasons for permanent discontinuation are:
* Condition under investigation resolved prior to minimum treatment period
* AE or any other condition posing a risk to a participant or jeopardizing safety
* Investigator, national coordinators, medical monitor, and/or Sponsor decided it is in the best interest of the participant's safety
* Positive pregnancy test during the treatment period
* Absence of explanation for liver injury and/or increase in liver function tests or acute kidney toxicity
* Discontinuation of intervention does not represent withdrawal from the study and participants should remain in the study until the end of the study (EOS).

ELIGIBILITY:
Inclusion Criteria

Participants must meet the following key inclusion criteria to be eligible for enrollment into the study:

1. Participants ≥9 months to <18 years of age at Screening; Female (post-menarchal) participants must have a negative serum/urine pregnancy test (β hCG sensitivity ≥25 mIU/mL).
2. Suspected/confirmed cIAI, cUTI, HAP/VAP, or BSI with gram-negative pathogens.
3. Require hospitalization and IV antibiotic treatment.

Exclusion Criteria

Participants with any of the following characteristics/conditions will be excluded:

1. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
2. Gram-negative species not expected to respond to ATM AVI ≤14 days.
3. Pregnant or breastfeeding; fertile male/female unwilling/unable to use effective contraception for at ≥7 days (males) or ≥28 days (females) after last ATM-AVI infusion.

   (HAP/VAP only):
4. Microbiologically known or high likelihood of monomicrobial infection with a gram-positive organism, lung abscess, pleural empyema, or post-obstructive pneumonia, lung or heart transplant.
5. Received >24 hours of systemic antibiotics during the 48 hours before randomization unless participant has documented treatment failure after at least 48 hours of antibiotic therapy.
6. Current use of any prohibited concomitant medication(s) or unwilling/unable (Cockayne Syndrome patients with cIAI are excluded) to use MTZ or having received previous investigational drug(s) or vaccine ≤30 days or 5 half-lives before randomization (whichever is longer).
7. CrCL ≤15 mL/min/1.73 m2 (eCrCl or eGFR calculation based on age).
8. Non-infectious related screening ALT or AST >3 x ULN, ALP >3 x ULN and/or TBili >2 x ULN (> 3 x ULN for Gilbert's syndrome).
9. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 9 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-08-17 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Maximum Predicted Plasma Concentration (Cmax) of ATM and AVI | Up to 15 Days
  Cmax is the maximum plasma concentration of ATM and AVI as population pharmacokinetic (popPK) analysis predicts.
Minimum Predicted Trough Plasma Concentration (Cmin) of ATM and AVI | Up to 15 Days
  Cmin is the minimum trough plasma concentration of ATM and AVI as popPK analysis predicts.
Area under the Concentration-Time Curve (AUC) of ATM-AVI | Up to 15 Days
  AUC is a measure of the plasma concentration of ATM and AVI overtime as popPK analysis predicts.
Plasma Decay Half-Life (t1/2) | Up to 15 Days
  Half-life is the time measured for the plasma concentration of ATM and AVI to decrease by one half as popPK analysis predicts.
Apparent Clearance (CL) | Up to 15 Days
  ATM and AVI clearance is a quantitative measure of the rate at which ATM and AVI are removed from the blood (rate at which ATM and AVI are metabolized or eliminated by normal biological processes). Clearance obtained after intravenous infusion dose (apparent clearance) is influenced by the fraction of the dose absorbed.
Proportion of Participants reporting Adverse Events (AE) | Baseline up to Day 50
  Proportion of participant AE reports of vital signs, physical examinations, and clinical laboratory tests overall and by age cohort. For each AE the last assessment made prior to the first dose of study drug will be defined as the baseline.
Proportion of Participants reporting Serious Adverse Events (SAE) | Baseline up to Day 50
  Proportion of participant SAE reports of vital signs, physical examinations, and clinical laboratory tests overall and by age cohort. For each SAE the last assessment made prior to the first dose of study drug will be defined as the baseline.
Proportion of Participants reporting AEs leading to discontinuation | Baseline up to Day 50
  Proportion of Participants reporting AEs leading to discontinuation from baseline. For each discontinuation the last assessment made prior to the first dose of study drug will be defined as the baseline
Proportion of Participants reporting AEs resulting in death | Baseline up to Day 50
  Proportion of Participants reporting AE resulting in death from baseline. For each death the last assessment made prior to the first dose of study drug will be defined as the baseline
Proportion of Participants reporting liver injury and acute kidney injury of ATM-AVI relative to Best Available Therapy (BAT) | Baseline up to Day 50
  Proportion of Participants reporting liver injury and acute kidney injury of ATM-AVI relative to Best Available Therapy (BAT) from baseline. For each report of liver and acute kidney injury the last assessment made prior to the first dose of study drug will be defined as the baseline

SECONDARY OUTCOMES:
Perentage of participants with favorable clinical response (CR) at end of iv study treatment (EOIV) | Up to 15 days after iv study drug treatment
  EOIV favorable CR is baseline signs and symptoms have improved such that with in 24hours after iv study treatment stopped, or premature discontinuation of the study drug or early withdrawal from the study no further antimicrobial treatment for the index infection is required. In addition, for cIAI participants, no unplanned drainage or surgical intervention is necessary since the initial procedure.
Percentage of Participants With Favorable Clinical Response (CR) at End of Treatment (EOT) | EOT within 48 hours after last dose of oral switch therapy or at time of premature discontinuation of study drug or early withdrawal from study
  EOT is only for those that were switched to oral therapy a favorable CR is baseline signs and symptoms have improved such that after study treatment, no further antimicrobial treatment for the index infection is required. In addition for cIAI participants, no unplanned drainage or surgical intervention is necessary since the initial procedure.
Percentage of Participants With Favorable Clinical Response (CR) at Test of Cure (TOC) | Up to 15 Days after last study treatment
  A TOC favorable CR is baseline signs and symptoms have improved such that after up to 14 days of study treatment, no further antimicrobial treatment for the index infection is required. In addition for cIAI participants, no unplanned drainage or surgical intervention is necessary since the initial procedure.
Percentage of participants with Favorable Microbiological Response at end of iv study drug treatment (EOIV) | EOIV within 24 hours after last iv study drug infusion
  Eradication (or urine quantification <103 CFU/mL for cUTI participants) of causative pathogen from an appropriately obtained specimen at the site of infection and presumed eradication specific to cIAI and HAP/VAP participants when repeat culture of specimens were not performed or clinically indicated in a participant who had a clinical response of cure
Percentage of Participants with Favorable Microbiological Response at End of Treatment (EOT) | EOT within 48 hours after last dose of oral switch therapy or at time of premature discontinuation of study drug or early withdrawal from study
  Eradication (or urine quantification <103 CFU/mL for cUTI participants) of causative pathogen from an appropriately obtained specimen at the site of infection and presumed eradication specific to cIAI and HAP/VAP participants when repeat culture of specimens were not performed or clinically indicated in a participant who had a clinical response of cure in participants who were switched to oral therapy
Percentage of Participants with Favorable Microbiological Response at test of cure (TOC) | Up to 15 Days
  Eradication (or urine quantification <103 CFU/mL for cUTI participants) of causative pathogen from an appropriately obtained specimen at the site of infection and presumed eradication specific to cIAI and HAP/VAP participants when repeat culture of specimens were not performed or clinically indicated in a participant who had a clinical response of cure.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (6):
  - Rady Children's Hospital, San Diego, California
  - Weill Cornell Medicine-New York Presbyterian Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Mount Sinai Kravis Children´s Hospital, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Le Bonheur Children's Hospital, Memphis, Tennessee
- China (3):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Shanghai Children's Medical Center, Shanghai
- Greece (2):
  - University General Hospital of Heraklion, Heraklion, Irakleío
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
- Semmelweis Egyetem, Budapest, Hungary
- India (5):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - RajaRajeswari Medical College and Hospital, Bangalore, Karnataka
  - Sahaydri Super Speciality Hospital, Nagar road, Pune, Maharashtra
  - Medanta Hospital Lucknow, Lucknow, Uttar Pradesh
  - Institute of Child Health, Kolkata, West Bengal
- Spain (6):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [barcelona]
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [barcelona]
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (3):
  - Hsinchu Municipal Mackay Children's Hospital, Hsinchu, Hsinchu
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (2):
  - Cukurova Universty, Sarçam, Adana
  - Istanbul Universitesi Istanbul Tıp Fakultesi Hastanesi, Istanbul, İ̇stanbul

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3601008